CLINICAL TRIAL: NCT01061086
Title: An Epidemiological Study of Acute Coronary Syndromes in The Greek Population
Brief Title: An Epidemiological Study of Acute Coronary Syndromes in The Greek Population. The TARGET Study
Acronym: TARGET
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Hellenic Cardiovascular Research Society (Other)
Responsible Party: Sponsor
Other Study IDs: NIS-CGR-DUM-2009/1
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Epidemiology; Management of disease; Outcomes; Greece
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients over 18 years old admitted to the hospital with Acute Coronary Syndrome.

SUMMARY:
This is a multicenter, 2-phase observational study of acute coronary syndromes (ACS) in Greece, designed to provide real world data on the risk factors of patients presenting to a hospital emergency department with an index event, as well as to depict the current management practices and outcomes of these clinical conditions in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an ACS (STEMI, NSTEMI, UA).
* Informed Consent

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff and staff at the study sites).
* Participation in other clinical study in period between the index event and 6- month follow-up assessment with the exception of registering in registries or surveys not influencing the management of the ACS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Room
Sampling Method: Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the proportion of patients who are on target for LDL-C according to the 2004-updated NCEP ATPIII guidelines as calculated within the first 24-hours of hospital admission for an ACS. | first visit - 1st day (cross-sectional part)
To estimate the proportion of patients enrolled in the cross-sectional part of the study that experiences a Major Adverse Cardiovascular Event (MACE) within a 6-month follow-up period. | follow up visit - 6th month (prospective part)

SECONDARY OUTCOMES:
To estimate the proportion of patients admitted to the hospital with STEMI, NSTEMI and unstable angina. | first visit - 1st day (cross-sectional part)
To estimate the "pain-to-door-time" throughout different regions in Greece. | first visit - 1st day (cross-sectional part)
To estimate the time to first MACE and to estimate CV, non-CV and all cause mortality within the 6-month period following the index ACS event. | follow up visit - 6th month (prospective part)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, Study Director — AstraZeneca
Locations (11):
- Greece (11):
  - Research Site, Athens, Attica
  - Research Site, Chalcis, Chalkida
  - Research Site, Chania, Chanion
  - Research Site, Chios, Chios
  - Research Site, Heraklion, Herakliou
  - Research Site, Ioannina, Ioanninon
  - Research Site, Ptolemaida, Kozani
  - Research Site, Larissa, Larrisis
  - Research Site, Volos, Magnisias
  - Research Site, Eddesa, Pella
  - Research Site, Komotini, Rodopi